CLINICAL TRIAL: NCT01457664
Title: A Randomized, Double-Blind, Multiple Dose, Placebo-Controlled, Study to Investigate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics of RO4995819 Following Oral Administration in Healthy Elderly Subjects.
Brief Title: A Study of RO4995819 in Healthy Elderly Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: BP25589
Record Dates: First submitted 2011-10-17; First posted 2011-10-24 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Healthy Volunteer

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- RO4995819 (Experimental)
  Interventions: Drug: RO4995819

INTERVENTIONS:
Drug: Placebo — Placebo to RO4995819 once daily for 14 days
  Arms: Placebo
Drug: RO4995819 — RO4995819 doses once daily for 14 days
  Arms: RO4995819

SUMMARY:
This study will evaluate the safety, tolerability and pharmacokinetics of RO4995819 in healthy elderly volunteers. Volunteers will be randomized to receive once daily doses of RO4995819 or matching placebo. The anticipated time on study treatment is 14 days.

ELIGIBILITY:
Inclusion Criteria:

* Adult healthy volunteer, 65-85 years of age
* Body Mass Index (BMI) between 18.0 to 30.0 kg/m2 inclusive and a total body weight >50 kg (110 lbs)
* Able to participate and willing to give written informed consent and to comply with the study restrictions

Exclusion Criteria:

* Any history or suspicion of drug or alcohol abuse
* Clinically significant or unstable cardiovascular or bronchopulmonary diseases, or any type of cancer
* History of liver disease
* Significant past or present neurological disorder
* History of psychiatric disorders
* Participation in an investigational drug or device study within 12 weeks prior to screening
* Donation of blood over 500 mL within three months prior to screening

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-07; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Safety (incidence of adverse events) | 8 weeks

SECONDARY OUTCOMES:
Pharmacokinetics: area under the concentration time curve (AUC) | Days 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, 16, 22, 20, 36, 62

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Miramar, Florida, United States